CLINICAL TRIAL: NCT05762718
Title: Validation of a Food Frequency Questionnaire: VioScreen
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 22-0904
Record Dates: First submitted 2023-02-22; First posted 2023-03-10 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2023-03

CONDITIONS: Not Determined

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to learn more about how well a questionnaire about food intake works. The study team will compare questionnaire responses to several other measurements of food intake. There is a special emphasis on fruit and vegetable intake.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 as we are aiming to recruit women of child-bearing age
* Pregnant women up to 26 weeks' gestation
* Women assigned female sex at birth who are not pregnant

Exclusion Criteria:

* Women below the age of 18 or over the age of 40 years
* Pregnant women more than 26 weeks' gestation at the time of enrollment
* Women who are experiencing limited or reduced food intake related to nausea will not be approached for recruitment and are considered ineligible
* Women who are unwilling to participate in the study due to time commitment or other reasons
* Women whose capacity for study compliance is diminished due to conditions such as active untreated substance use disorder, untreated/uncontrolled schizophrenia, bipolar disorder, active psychosis will not be approached for recruitment and are considered ineligible

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women of child-bearing age
Study Population: pregnant women and women of child-bearing age
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Concurrent validity of VioScreen against 24-hour recalls | 6 weeks
  Concurrent validity measures how a new test compares against a validated test, called the criterion or "gold standard."
Test-retest reliability of VioScreen | one month
  Test-retest reliability is a measure of reliability obtained by administering the same test twice over a period of time to a group of individuals.

SECONDARY OUTCOMES:
Concurrent validity of VioScreen against Veggie Meter | 6 weeks
  Concurrent validity measures how a new test compares against a validated test, called the criterion or "gold standard."
Concurrent validity of VioScreen against Fruit and Vegetable Screener | 6 weeks
  Concurrent validity measures how a new test compares against a validated test, called the criterion or "gold standard."
Test-retest reliability of Veggie Meter | one month
  Test-retest reliability is a measure of reliability obtained by administering the same test twice over a period of time to a group of individuals.
Test-retest reliability of Fruit and Vegetable Screener | one month
  Test-retest reliability is a measure of reliability obtained by administering the same test twice over a period of time to a group of individuals.
Concurrent validity of Veggie Meter against 24-hour recalls | 6 weeks
  Concurrent validity measures how a new test compares against a validated test, called the criterion or "gold standard."
Concurrent validity of Fruit and Vegetable Screener against 24-hour recalls | 6 weeks
  Concurrent validity measures how a new test compares against a validated test, called the criterion or "gold standard."

CONTACTS AND LOCATIONS:
Overall Officials: Carina Venter, PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Children's Hospital Colorado, Aurora, Colorado
  - Denver Health, Denver, Colorado